CLINICAL TRIAL: NCT07126873
Title: A Phase 1/2a Study to Evaluate the Safety, Tolerability, and Efficacy of E-islet 01 in Subjects Who Have Type 1 Diabetes Mellitus With Impaired Hypoglycemic Awareness and Severe Hypoglycemia
Brief Title: A Safety, Tolerability, and Efficacy Study of E-islet 01 in Participants With Type 1 Diabetes
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: EndoCell Therapeutics, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ENDOCELL-T1DM-101
Record Dates: First submitted 2025-08-10; First posted 2025-08-17 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Diabetes Mellitus, Type 1; Impaired Hypoglycemic Awareness; Severe Hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Allogeneic Human E-islet (E-islet 01) (Experimental)
  Interventions: Biological: Allogeneic Human E-islet (E-islet 01)

INTERVENTIONS:
Biological: Allogeneic Human E-islet (E-islet 01) — Allogeneic Human E-islet (E-islet 01), Infused into the hepatic portal vein

SUMMARY:
This study will evaluate the safety, tolerability and efficacy of E-islet 01 in participants with Type 1 diabetes mellitus (T1D) and impaired awareness of hypoglycemia (IAH) and severe hypoglycemia

ELIGIBILITY:
Inclusion Criteria:

* Clinical history of Type 1 Diabetes with > 5 years of duration
* 2-hour C-peptide level <0.3 ng/mL after a mixed meal stimulation test
* Under continuous insulin therapy, Participants have at least one of the following conditions:

  1. At least one episode of documented severe hypoglycemia in the 12 months prior to enrollment;
  2. Unaware hypoglycemia evaluated using the Clarke scoring system
* Willing and able to conduct self-blood glucose monitoring as required, with good compliance
* Voluntarily participate and sign the informed consent form

Exclusion Criteria:

* Uncontrolled systemic infections, including but not limited to pulmonary tuberculosis, active hepatitis, a history of positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV-Ab), human immunodeficiency virus antibody (HIV-Ab), or Treponema pallidum antibody (TP-Ab).
* History of malignancy within the past 5 years or undergoing antitumor treatment
* Participation in other clinical trials in the 3 months or islet cell transplant, organ transplant, or cell therapy in the 12 months prior to enrollment
* Other situations judged by the investigator as unsuitable for participation in the trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-08-11 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From E-islet 01 infusion to end of study (up to 5 years)
Proportion of Participants Free of Severe Hypoglycemic Events With Either a Glycated Haemoglobin (HbA1c) <7.0% or a ≥ 1% Reduction in Glycosylated hemoglobin(HbA1c) From Baseline | At 1 year after E-islet 01 infusion

SECONDARY OUTCOMES:
Proportion of Participants who are Time in range (TIR) >70% | At 1 year after E-islet 01 infusion
Number of participants with increase in fasting C-peptide and stimulated C-peptide from baseline | At 1 year after E-islet 01 infusion
Proportion of Participants who are Insulin Independent or Reduction in Exogenous Insulin | At 1 year after E-islet 01 infusion

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China